CLINICAL TRIAL: NCT05203003
Title: Prospective Evaluation of the Prognostic Impact of Measurable Residual Disease (MRD) Within a Phase III Study Comparing a Fixed Duration Therapy Versus Continuous Therapy With Daratumumab, Lenalidomide, and Dexamethasone for Relapsed Multiple Myeloma Requiring a First Salvage Treatment.
Acronym: MRD-CONFIRM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210482
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; measurable residual disease; daratumumab; lenalidomide; dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients who are included in the CONFIRM phase III trial
  Interventions: Other: Assessment of MRD

INTERVENTIONS:
Other: Assessment of MRD — Bone marrow aspirate for assessment of MRD will be performed at 2 years (+/- 3 month) after randomization in patients still under treatment and in complete response.
  Thereafter, bone marrow aspirate for assessment of MRD will be repeated at 3 and 4 years in patients that maintain complete response, irrespective of the randomization arm and therefore of treatment administration.

SUMMARY:
We propose to conduct an ancillary prospective evaluation of the impact of Dara-Len-Dex discontinuation after 2 years, on the persistence of MRD negativity in patients that were MRD negative at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) who are included in the CONFIRM phase III trial (ClinicalTrials.gov Identifier: NCT03836014).
* Subject that are still under therapy at 2 years (+/- 3 month) after randomization, either in the fixed duration therapy group or in the continuous therapy group of the CONFIRM protocol
* Subject in complete response at 2 years (+/- 3 month) after randomization.
* Signed informed consent
* Affiliation to a social security system or equivalent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are included in the CONFIRM phase III trial
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients that maintain MRD negativity | 3 and 4 years after inclusion
  Rate of patients that maintain MRD negativity at 3 and 4 years after inclusion in the current protocol in the continuous Dara-Len-Dex therapy group versus fixed duration Dara-Len-Dex therapy (2 years) group.

SECONDARY OUTCOMES:
PFS at 2 years | 2 years
  PFS at 2 years after initial assessment of MRD negativity, which is defined as the duration from the date of MRD measurement to either progressive disease, according to the IMWG criteria, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Hematology, Hospital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No